CLINICAL TRIAL: NCT04758754
Title: Active and Passive Exercise Training in Improving Vascular Function: Local vs Systemic Vascular Effect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Universita di Verona (Other)
Responsible Party: Principal Investigator, Emilano Cè, Associate Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Active vs passive training
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Aerobic Exercise; Stretching

STUDY DESIGN:
Intervention Model Description: Three arms: 1) active exercise training (single leg knee extension); 2) passive exercise training (passive static training); 3) controls (no training)
Who Masked: Outcomes Assessor
Masking Description: Blind to intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single leg knee extension training (SLKE) (Experimental): Active 8-week training involving lower limbs. SLKE participants will be involved in a 8-week aerobic training protocol involving the knee extensor muscles. The training will be held on an Anderson and Saltin ergometer, 3 times per week, with a single session duration of 33.3 min. Total weekly duration: 100 min.
  Interventions: Other: Training
- Passive static stretching training (PST) (Active Comparator): Passive 8-week training involving lower limbs. PST participants will be involved in a 8-week passive static training training involving the knee extensor muscles. The training will have a frequency of 5 times per week, with a single duration of 20 min. Total weekly duration: 100 min
  Interventions: Other: Training
- Control (CTRL) (No Intervention): CTRL will not receive any intervention.

INTERVENTIONS:
Other: Training — 8-weeks iso-volume active (SLKE) or passive static stretching training (PST) involving lower limb muscles
  Arms: Passive static stretching training (PST); Single leg knee extension training (SLKE)

SUMMARY:
Maintaining an adequate state of vascular function is an important element for the maintenance of cardiovascular well-being. Several training plans involving both active and passive engagement by the muscles have been proposed with the aim of improving vascular function. At local level, i.e., at the level of the arteries that supply the muscles directly involved in training, significant improvements in vascular function have been found. These improvements are more noticeable after active training than with a passive training regimen, such as passive static stretching. On the contrary, at the systemic level the effects of active or passive training are less clear and, above all, it is not evident whether there is a difference in the effects induced at the level of vascular function in arteries supplying muscles not directly involved in training. The aim of the study is to clarify the local and systemic effect of an active training protocol (single leg knee extension, SLKE) and of a passive training protocol (passive static stretching training, PST) applied to the lower limbs lasting 8 weeks on the local (femoral artery) and systemic (brachial artery) vascular function.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* neurological, vascular and musculoskeletal disorders of the lower and upper limbs;
* being on pharmacological therapy related to either neural and/or vascular response, including hormonal contraceptives and oral supplements;
* being a current or former smoker;
* having an irregular menstrual cycle (26 to 35 days) up to 3 months before the beginning of the study;
* contraindications to joint mobilization; regular involvement in a SLKE or PS training programme.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in brachial artery flow mediated dilation | Change from baseline in percentage flow mediated dilation at 8 weeks
  Flow mediated dilation was performed at brachial artery level. An arterial pressure cuff was placed around the forearm immediately distal to the olecranon process to provide an ischemic stimulus when inflated. Following baseline assessment, the blood pressure cuff was inflated to 250 mmHg. Artery diameter was and blood flow were resumed at baseline, 30 s prior to cuff deflation and continued for 2 min post-deflation by a linear array transducer attached to a high-resolution ultrasound machine. When an optimal image was obtained, the probe was held stable and longitudinal in B-mode, acquiring images of the lumen-arterial wall interface. Continuous Doppler velocity assessments were also obtained and collected using the lowest possible insonation angle (<60°). Data were exported and analyzed using commercially available software. Flow mediated dilation was quantified as the maximal change in artery diameter after cuff release, expressed as a percentage increase above baseline (%).

SECONDARY OUTCOMES:
Change from baseline in femoral artery delta blood flow | Change from baseline in Delta Blood Flow at 8 weeks
  Femoral artery blood flow was calculated by Doppler ultrasound at baseline and at peak after single passive knee flexion and extension by using the femoral artery diameter and mean blood velocity. The difference between baseline and at peak blood flow identifies the Delta Blood Flow (ml/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Science for Health, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Statistical Analysis Plan
Supporting Information: Study Protocol, SAP
Time Frame: Data publication up to three years from publication
Access Criteria: Mail to Corresponding Author

REFERENCES:
- [Derived] Ce E, Venturelli M, Bisconti AV, Longo S, Pedrinolla A, Coratella G, Schena F, Esposito F. Long-Term Passive Leg Stretch Improves Systemic Vascular Responsiveness as Much as Single-Leg Exercise Training. Med Sci Sports Exerc. 2022 Mar 1;54(3):475-488. doi: 10.1249/MSS.0000000000002811. PMID 34690287